CLINICAL TRIAL: NCT02177370
Title: Effect of Fenoterol Metered Dose Inhaler (0.1 mg) on the Beta-receptor Population on Lymphocytes and the Clinical Findings Compared With Treatment With DSCG Metered Dose Inhaler in Patients With Bronchial Asthma.
Brief Title: Effect on Fenoterol Metered Dose Inhaler on the Beta-receptor Population on Lymphocytes in Patients With Bronchial Asthma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 260.716
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (2):
- Fenoterol metered dose inhaler (MDI) (Experimental)
  Interventions: Drug: Fenoterol MDI
- DSCG MDI (Active Comparator)
  Interventions: Drug: DSCG MDI

INTERVENTIONS:
Drug: Fenoterol MDI
  Arms: Fenoterol metered dose inhaler (MDI)
Drug: DSCG MDI
  Arms: DSCG MDI

SUMMARY:
The aim of the study was to compare the effect of fenoterol metered dose inhaler with disodium cromoglycate (DSCG) metered dose inhaler on the lymphocyte β2-receptor population as well as on the clinical findings in patients with bronchial asthma over a two-week period of treatment.

ELIGIBILITY:
Inclusion Criteria:

* sex: male and female
* age: 18 years or over
* bronchial asthma, diagnosis confirmed by history and positive inhalation challenge test (unspecific challenge with carbachol, PD100SRaw))
* severity of asthma mild to moderate or asthmatic in symptom-free intervals
* Raw ≤ 5 cm H2O/l/s
* no antiasthmatic treatment in the week (steroid therapy: two weeks) before the start of the study

Exclusion Criteria:

* clinically significant, concomitant haematological, cardiac, renal, hepatic or metabolic diseases
* intercurrent diseases, e.g. severe respiratory infections
* patients who cannot do without the following preparations during the 5-week trial:

  * inhaled/oral steroids
  * theophylline
  * antihistamine, antiallergic drugs
  * inhaled/oral sympathomimetics
  * anticholinergics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1990-02; Primary Completion 1996-10 (Actual)

PRIMARY OUTCOMES:
Airway resistance (Raw) | after 2 weeks
Number of binding sites of the β2 receptors per lymphocytes (BS/LY) | after 2 weeks